CLINICAL TRIAL: NCT06721728
Title: Effect of Oral Health Educational Program on the Oral Health-Related Quality of Life of a Group of Children With Type-1 Diabetes Mellitus: A Before and After Pilot Study
Brief Title: Effect of Oral Health Educational Program on Oral Health Quality of Life of Group of Type1 Diabetes Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farida Mohsen Abd El Satar, dentist, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CEBD-CU-2024-11-07
Record Dates: First submitted 2024-11-27; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Oral Health Related Quality of Life

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Type 1 diabetes mellitus children (Experimental): children diagnosed with type 1 diabetes mellitus will receive an educational program with oral hygiene measures and diet advice related to their condition.
  Interventions: Behavioral: Oral health educational program

INTERVENTIONS:
Behavioral: Oral health educational program — Flyer distributed on the children with data about oral hygiene measures as well as diet advice related to their condition, in addition to modeling the correct tooth brushing habits using a cast and tooth brush.

SUMMARY:
The study is a before and after study made to assess the oral health related quality of life after oral health educational program on children with type1 diabetes mellitus.

The main questions it aims to answer are:

* oral health related quality of life
* caries experience

Participants will answer oral health quality of life questionnaire and will be checked for DMF and def indices and then given an oral health education program and followed up after 3 months.

DETAILED DESCRIPTION:
The oral health educational program will be conducted in Arabic in the form of flyers given to the children and their parents plus modeling on brushing habits on a cast and tooth brush.The educational program will emphasize on three main messages (brushing twice daily, healthy diet compatible with their disease and regular dentist visits).

Data in the flyer contained dietary tips as well as oral hygiene habits, design was made by the primary investigator.

The child oral health related quality of life will be measured by the validated Arabic child perception questionnaire (CPQ8-10)

Dental history, def and DMF indices will be measured by dental chart that will be modified to include a section for current medications.

To avoid selection bias all participants matching inclusion criteria in examination day will be included and all outcomes will be reported to avoid reporting and detection bias.

Study size: To the best of our knowledge there are no other studies found in literature to estimate a sample size so this study is going to be a pilot study with sample size of 50 child.

Statistical method: Categorical data will be represented as frequency (n) and percentage (%) and will be analyzed using chi square test. Numerical data will be investigated for normality by checking the data distribution, calculating the mean and median values and using Kolmogorov-Smirnov and Shapiro-Wilk tests. If the data was normally distributed, it will be shown as mean and standard deviation values and an independent t-test will be used for analysis. If the assumption of normality was violated; the data will be presented as median and range values and will be analyzed using Mann-Whitney U test. The significance level will be set at p ≤0.05 for all tests. Statistical analysis will be performed with IBM® SPSS® Statistics Version 26 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes
* Age from 8 to 10 years old
* Diagnosed with type 1 diabetes mellitus

Exclusion Criteria:

* Children with other systemic diseases
* Parents who refuse participation

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
oral health related quality of life | Measured before the educational program and then after 3 months from receiving the educational program
  change in oral health related quality of life before and after the educational program measured in percentage

SECONDARY OUTCOMES:
caries experience | Measured before the educational program and then after 3 months from receiving the educational program
  Caries experience will be measured using DMF and def indices before and after the educational program and will be represented by mean and standard deviation